CLINICAL TRIAL: NCT06836362
Title: Acupuncture for Children with Functional Constipation: a Pilot Study
Brief Title: Acupuncture for Children with Functional Constipation
Acronym: ACU-PILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.A. Benninga, Prof. Dr. M.A. Benninga, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL87083.018.24
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Functional Constipation (FC)
Keywords: functional constipation; child; acupuncture; children; DGBI; pilot study
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm study. The intervention consists of acupuncture treatments (Other): This is an open-label, non-randomized single-arm study. The intervention consists of acupuncture (see description under intervention). Throughout the study duration, participants will maintain their therapeutic recommendations related to treating constipation (PEG at the dosage prior to entering the study, minimum of 0.2 g/kg/day, education and non-pharmacological advice as previously described by the medical team in charge). Initiation of new treatments for FC or increasing the dosage of PEG is not allowed during the intervention period. Decreasing the dosage of PEG is allowed if instructed by the treating physician and will be documented. After the last acupuncture session, if the patient requires an increase in the dosage of PEG, this is allowed during the follow-up period and will be documented. As per current treatment guidelines, participants are allowed to use escape medication (bisacodyl or enemas) after 72 hours without defecation or when their symptoms become intolerable.
  Interventions: Other: Acupuncture treatment

INTERVENTIONS:
Other: Acupuncture treatment — Children will receive 8 acupuncture sessions during 10 weeks (1 session per week during 6 weeks, followed by 1 session every other week during 4 weeks).
  At each acupuncture session, the acupuncturist records the patient's bowel habits, gastrointestinal symptoms and the use of escape medication during the period between sessions. After 3, 6 and 8 acupuncture treatments respectively, patients will visit the research team after they receive acupuncture to evaluate adverse events.
  After completion of these 10 weeks, an acupuncture-free follow-up period of 4 weeks commences. The follow-up period will be used to investigate if and how long effects of the intervention will persist. During the intervention period and the follow-up period, escape medication (bisacodyl or enemas) is allowed under the same conditions as during the run-in period.

SUMMARY:
Background of the study:

Functional constipation (FC) is common in children and poses a significant burden to patients, their families and the healthcare system. Pharmacological treatment mainly consists of oral osmotic laxatives. However, poor adherence to oral laxatives is known to be a common problem and patients often remain symptomatic despite pharmacological treatment. Many parents seek help in the form of complementary and integrative medicine. Acupuncture has been shown to relieve symptoms in adults with FC. However, published studies in children with FC are scarce and have important limitations.

Objective of the study:

To evaluate the feasibility, safety and potential efficacy of acupuncture in children with FC. The results of this study will be used to design a future randomized controlled trial (RCT).

Study design:

A prospective, non-randomized, multicenter, open-label pilot study.

Intervention: Children will receive 8 acupuncture sessions during 10 weeks (1 session per week during 6 weeks, followed by 1 session every other week during 4 weeks). Concurrent pharmacological treatment with polyethylene glycol ≥ 0.2 g/kg/day will be maintained as initiated prior to participation in the study.

Study population:

18 children (6-18 years old) with FC according to the Rome IV criteria.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:
* 6-18 years of age
* meet the modified Rome IV criteria for FC (defined as meeting at least two of the following criteria during the 2-week run-in period despite receiving treatment with PEG with a minimum dose of 0.2 g/kg/day):

  1. Two or fewer spontaneous bowel movements (SBMs) per week (an SBM is defined as a bowel movement that occurs in the absence of laxative, enema, or suppository use in the preceding 24 hours)
  2. History of excessive stool retention
  3. History of painful or hard bowel movements
  4. History of large-diameter stools
  5. Presence of a large fecal mass in the rectum
  6. At least 1 episode/week of incontinence after the acquisition of toileting skills
  7. History of large-diameter stools that may obstruct the toilet in toilet-trained children
* Insufficient symptom management despite at least three months of medical management (including education, non-pharmacological advice and laxatives) by a physician. Insufficient symptom management is defined as the presence of at least one of the Rome IV criteria for FC despite medical management by a physician.
* are treated with PEG with a minimum dose of 0.2 g/kg/day for a minimum of 1 month prior to inclusion in the study
* Written informed consent obtained from parents or guardians and all children ≥12 years.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* children with FC not treated with PEG with a minimum dose of 0.2g/kg/day during at least one month at the time of potential inclusion.
* Irritable bowel syndrome.
* Organic causes of constipation; e.g. celiac disease, pediatric intestinal pseudo-obstruction, hypothyroidism, spina bifida, anorectal malformations, or Hirschsprung disease.
* Significant chronic health conditions requiring specialty care (e.g. cardiac, pulmonary, hepatic, hematopoietic, renal, endocrine, or metabolic diseases, sickle cell disease, cerebral palsy) that could potentially impact the child's ability to participate or confound the results of the study.
* Unintentional weight loss greater than or equal to 5% of their body weight within the last 3 months.
* Gastrointestinal blood loss.
* Recurrent or unexplained fevers.
* Pregnancy.
* Smoking.
* History of abdominal surgery involving the luminal gastrointestinal tract, except appendectomy or hernia repairs.
* Concomitant use of drugs that are known to affect gastrointestinal motility.
* Established diagnoses of autism spectrum disorders.
* Major psychiatric disorders (bipolar disorder, schizophrenia, major depression) or a history of abuse.
* Severe needle-related anxiety.
* Rash or active local infection over an acupuncture point.
* Immunocompromised children (specifically inadequately regulated diabetes mellitus, active staphylococcal-related skin conditions)
* Clotting disorders or a recent history of thrombocytopenia.
* Children who previously received acupuncture for constipation.
* Children who currently participate in another clinical trial.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure: feasibility | From enrollment until the end of the intervention period (at 10 weeks)
  The primary endpoint is feasibility: a future RCT using this same intervention protocol will be deemed feasible if the pilot study renders an attrition rate ≥70% (i.e. ≥70% of patients completing the pilot study while attending ≥75% of scheduled acupuncture sessions).

SECONDARY OUTCOMES:
Secondary outcome measure: Feasibility | From enrollment to the end of intervention (week 10) and follow-up (week 14)
  Secondary endpoints to determine feasibility include consent rate, patient and parent satisfaction with acupuncture treatment (measured at t=6, t=10 and t=14 [5-point-Likert scale]) and assessment of required personnel capacity for a future RCT
Secondary Outcome Measure: Safety (assessment of adverse events) | From first acupuncture treatment until last treatment (week 10) and after follow-up (week 14)
  The occurrence of adverse events (AE) is assessed at each research nurse visit (t=3, t=6, t=10, t=14). The occurrence of the following pre-determined adverse events are assessed: needle-related pain, local redness/irritation, hematomas, headache, fainting/syncope, sedation, neuropathy. For each patient-reported AE, severity (mild, moderate, or severe) and relation to acupuncture treatment (unrelated or possibly, probably, or definitely related) are determined.
Secondary Outcome Measure: Efficacy | From start of intervention until end of intervention (at week 10 and at follow-up (at week 14)
  The endpoint for efficacy is treatment success, based on the Rome IV criteria (Table 1): a child who fulfils the Rome IV criteria for FC prior to enrolment into the trial and no longer fulfils the Rome IV criteria at the end of the trial period is considered successfully treated. The endpoints, including quality of life and school absence, are based on a previously published core outcome set and include:
  * Defecation frequency (number of bowel movements/week, excluding fecal incontinence episodes)
  * Stool consistency (Bristol Stool Scale)
  * Painful defecation (yes/no)
  * Fecal incontinence frequency (episodes/week)
  * Withholding behavior (yes/no)
  * Abdominal pain (yes/no, VAS score)
  * Number of spontaneous bowel movements (>24h after escape medication)
  * Time between acupuncture and defecation
  * Number of bowel movements <24h after acupuncture
  * Frequency of use of escape medication
  * Time between escape medication and defecation
  * Number of bowel movements <24h after escape med.

REFERENCES:
- [Derived] Bloem MN, Baaleman DF, Koppen IJN, Vlieger AM, de Lorijn F, Birch S, Nieuwdorp M, Benninga MA. Prospective, non-randomised, open-label pilot trial assessing feasibility, safety and treatment success of acupuncture in children with functional constipation: ACU-PILOT study protocol. BMJ Open. 2025 Nov 11;15(11):e109425. doi: 10.1136/bmjopen-2025-109425. PMID 41218934